CLINICAL TRIAL: NCT04125459
Title: Assessing the Role of the NLRP3 Inflammasome in Driving Inflammation in Affected Joints of Patients With Intercritical Gout
Brief Title: Assessing the Role of the NLRP3 Inflammasome in Intercritical Gout
Status: Active, not recruiting | Type: Observational
Sponsor: Attune Health Research, Inc. (Industry)
Collaborators: Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Responsible Party: Principal Investigator, Swamy Venuturupalli, Founder of Attune Health, Attending Rheumatologist at Cedar Sinai Medical Center, Associate Clinical Professor of Medicine at UCLA, Attune Health Research, Inc.
Other Study IDs: 36549
Record Dates: First submitted 2019-09-23; First posted 2019-10-14 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The types of biospecimen collected will be 3-8 synovial tissue samples (from the ultrasound-guided synovial biopsy), as well as 60 mL of peripheral blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Gout: This arm will be getting a biopsy as well as a blood draw
  Interventions: Procedure: Joint Biopsy
- Controls: These individuals will not be getting a joint biopsy and will just get a blood draw

INTERVENTIONS:
Procedure: Joint Biopsy — a synovial biopsy of a joint that has been affected by a gout attack
  Groups: Individuals with Gout

SUMMARY:
Gout is an autoinflammatory disease characterized by flares of painful joint inflammation. This inflammation occurs in response to uric acid that crystallizes. After a gout attack, patients usually enter a period that is accompanied by low grade inflammation but is otherwise relatively asymptomatic. Gout is typically associated with certain markers, and this study is going describe specific markers in patients that are in between gout attacks. Research has been focused on studying this phase between gout attacks in hopes to manage and prevent the onset of future gout attacks. Biopsies will be taken from the affected joint and blood will be drawn from patients who are currently in between gout attacks. This work will provide important information regarding how crystals in the joint lining are associated with chronic inflammation in the periods between gout attacks. Moreover, this study will identify novel biomarkers that may be useful in determining the severity of disease activity through a blood test.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with gout diagnosed by a Rheumatologist.
2. patients with a history of at least two gout attacks in the target joint
3. Patients with a target joint amenable to biopsy. Target joint defined as:

Joint that has been affected by acute gout attack at least twice in the 12 months prior to enrollment.

Ultrasound finds grade 2 gray-scale synovitis in joint. Joint is amenable to biopsy. At the time of enrollment, the joint is without signs of acute inflammation: redness, swelling, and severe pain (>7/10).

Exclusion Criteria:

1. Patients on anti-coagulation therapy.
2. Patients with an active infection.
3. Tophus present at the biopsy site.
4. Target joint with signs of acute gout attack (pain >7/10, redness, warmth)
5. Known chondrocalcinosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients over the age of 18 diagnosed with intercritical gout who have evidence of inflammation as determined by ultrasound examination will be screened for this study. The control group will comprise of age and sex-matched healthy volunteers. They will be recruited from the private rheumatology practices of Swamy Venuturupalli, MD and Ami Ben-Artzi, MD.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2024-10-03 (Estimated)

PRIMARY OUTCOMES:
NLRP3 Inflammasome Role in Driving Inflammation in Intercritical Gout | Up to 2 months
  To investigate the role of the NLRP3 inflammasome in driving inflammation in intercritical gout. Specifically, this will be accomplished via measuring caspase-1 activity as a marker of inflammasome activity. We will measure the % of patients who show a %positivity (physiological parameter) of caspase-1 activity.
IL-1B Role in Driving Inflammation in Intercritical Gout | Up to 2 months
  Examine the role of IL-1b in driving inflammation within intercritical gout via the measurement of IL-1b levels. IL-1b concentration levels (physiological parameter) will be measured in ng/ml.

SECONDARY OUTCOMES:
Microcrystal Correlation | Up to 2 months
  Correlate NLRP3 activity with the presence of microcrystals in the synovium
Immune Cell Infiltration in the Inflamed Joint Correlation | Up to 2 months
  Correlate NLRP3 activity with the presence of infiltration of immune cells in the inflamed joint as determined by flow cytometry and cytology
Uric Acid Levels Correlation | Up to 2 months
  Correlate NLRP3 activity with the concentration of uric acid levels in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Swamy Venuturupalli, MD, Principal Investigator — Attune Health
Locations (1):
- Attune Health Research Inc., Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawrence RC, Helmick CG, Arnett FC, Deyo RA, Felson DT, Giannini EH, Heyse SP, Hirsch R, Hochberg MC, Hunder GG, Liang MH, Pillemer SR, Steen VD, Wolfe F. Estimates of the prevalence of arthritis and selected musculoskeletal disorders in the United States. Arthritis Rheum. 1998 May;41(5):778-99. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-V. PMID 9588729
- [Background] Zhu Y, Pandya BJ, Choi HK. Prevalence of gout and hyperuricemia in the US general population: the National Health and Nutrition Examination Survey 2007-2008. Arthritis Rheum. 2011 Oct;63(10):3136-41. doi: 10.1002/art.30520. PMID 21800283
- [Background] Neogi T, Hunter DJ, Chaisson CE, Allensworth-Davies D, Zhang Y. Frequency and predictors of inappropriate management of recurrent gout attacks in a longitudinal study. J Rheumatol. 2006 Jan;33(1):104-9. Epub 2005 Nov 1. PMID 16267879
- [Background] Burns CM, Wortmann RL. Latest evidence on gout management: what the clinician needs to know. Ther Adv Chronic Dis. 2012 Nov;3(6):271-86. doi: 10.1177/2040622312462056. PMID 23342241
- [Background] Ragab G, Elshahaly M, Bardin T. Gout: An old disease in new perspective - A review. J Adv Res. 2017 Sep;8(5):495-511. doi: 10.1016/j.jare.2017.04.008. Epub 2017 May 10. PMID 28748116
- [Background] Hirsch JD, Terkeltaub R, Khanna D, Singh J, Sarkin A, Shieh M, Kavanaugh A, Lee SJ. Gout disease-specific quality of life and the association with gout characteristics. Patient Relat Outcome Meas. 2010 Mar 1;2010:1-8. doi: 10.2147/PROM.S8310. PMID 21686040
- [Background] Pascual E. Persistence of monosodium urate crystals and low-grade inflammation in the synovial fluid of patients with untreated gout. Arthritis Rheum. 1991 Feb;34(2):141-5. doi: 10.1002/art.1780340203. PMID 1994910
- [Background] Carter JD, Patelli M, Anderson SR, Prakash N, Rodriquez EJ, Bateman H, Sterrett A, Valeriano J, Ricca LR. An MRI assessment of chronic synovial-based inflammation in gout and its correlation with serum urate levels. Clin Rheumatol. 2015 Feb;34(2):345-51. doi: 10.1007/s10067-014-2644-9. Epub 2014 May 7. PMID 24797771
- [Background] Ruggiero C, Cherubini A, Ble A, Bos AJ, Maggio M, Dixit VD, Lauretani F, Bandinelli S, Senin U, Ferrucci L. Uric acid and inflammatory markers. Eur Heart J. 2006 May;27(10):1174-81. doi: 10.1093/eurheartj/ehi879. Epub 2006 Apr 12. PMID 16611671
- [Background] Grainger R, McLaughlin RJ, Harrison AA, Harper JL. Hyperuricaemia elevates circulating CCL2 levels and primes monocyte trafficking in subjects with inter-critical gout. Rheumatology (Oxford). 2013 Jun;52(6):1018-21. doi: 10.1093/rheumatology/kes326. Epub 2012 Nov 30. PMID 23204548
- [Background] Kingsbury SR, Conaghan PG, McDermott MF. The role of the NLRP3 inflammasome in gout. J Inflamm Res. 2011;4:39-49. doi: 10.2147/JIR.S11330. Epub 2011 Mar 13. PMID 22096368
- [Background] Landis RC, Haskard DO. Pathogenesis of crystal-induced inflammation. Curr Rheumatol Rep. 2001 Feb;3(1):36-41. doi: 10.1007/s11926-001-0049-7. PMID 11177769
- [Background] Amaral FA, Costa VV, Tavares LD, Sachs D, Coelho FM, Fagundes CT, Soriani FM, Silveira TN, Cunha LD, Zamboni DS, Quesniaux V, Peres RS, Cunha TM, Cunha FQ, Ryffel B, Souza DG, Teixeira MM. NLRP3 inflammasome-mediated neutrophil recruitment and hypernociception depend on leukotriene B(4) in a murine model of gout. Arthritis Rheum. 2012 Feb;64(2):474-84. doi: 10.1002/art.33355. PMID 21952942
- [Background] Guo H, Callaway JB, Ting JP. Inflammasomes: mechanism of action, role in disease, and therapeutics. Nat Med. 2015 Jul;21(7):677-87. doi: 10.1038/nm.3893. Epub 2015 Jun 29. PMID 26121197
- [Background] Krishnan E, Baker JF, Furst DE, Schumacher HR. Gout and the risk of acute myocardial infarction. Arthritis Rheum. 2006 Aug;54(8):2688-96. doi: 10.1002/art.22014. PMID 16871533
- [Background] Jarrah AA, Tarzami ST. The duality of chemokines in heart failure. Expert Rev Clin Immunol. 2015 Apr;11(4):523-36. doi: 10.1586/1744666X.2015.1024658. Epub 2015 Mar 12. PMID 25764001
- [Background] Woollard KJ, Geissmann F. Monocytes in atherosclerosis: subsets and functions. Nat Rev Cardiol. 2010 Feb;7(2):77-86. doi: 10.1038/nrcardio.2009.228. Epub 2010 Jan 12. PMID 20065951
- [Background] Kuo CF, See LC, Luo SF, Ko YS, Lin YS, Hwang JS, Lin CM, Chen HW, Yu KH. Gout: an independent risk factor for all-cause and cardiovascular mortality. Rheumatology (Oxford). 2010 Jan;49(1):141-6. doi: 10.1093/rheumatology/kep364. Epub 2009 Nov 20. PMID 19933595
- [Background] Goldenberg DL, Cohen AS. Synovial membrane histopathology in the differential diagnosis of rheumatoid arthritis, gout, pseudogout, systemic lupus erythematosus, infectious arthritis and degenerative joint disease. Medicine (Baltimore). 1978 May;57(3):239-52. doi: 10.1097/00005792-197805000-00004. PMID 642792
- [Background] Agudelo CA, Schumacher HR. The synovitis of acute gouty arthritis. A light and electron microscopic study. Hum Pathol. 1973 Jun;4(2):265-79. doi: 10.1016/s0046-8177(73)80013-9. No abstract available. PMID 4350339
- [Background] Najm A, Orr C, Heymann MF, Bart G, Veale DJ, Le Goff B. Success Rate and Utility of Ultrasound-guided Synovial Biopsies in Clinical Practice. J Rheumatol. 2016 Dec;43(12):2113-2119. doi: 10.3899/jrheum.151441. Epub 2016 Oct 15. PMID 27744399
- [Background] Kelly S, Humby F, Filer A, Ng N, Di Cicco M, Hands RE, Rocher V, Bombardieri M, D'Agostino MA, McInnes IB, Buckley CD, Taylor PC, Pitzalis C. Ultrasound-guided synovial biopsy: a safe, well-tolerated and reliable technique for obtaining high-quality synovial tissue from both large and small joints in early arthritis patients. Ann Rheum Dis. 2015 Mar;74(3):611-7. doi: 10.1136/annrheumdis-2013-204603. Epub 2013 Dec 13. PMID 24336336
- [Background] Humby F, Kelly S, Hands R, Rocher V, DiCicco M, Ng N, Zou L, Bugatti S, Manzo A, Caporali R, Montecucco C, Bombardieri M, Pitzalis C. Use of ultrasound-guided small joint biopsy to evaluate the histopathologic response to rheumatoid arthritis therapy: recommendations for application to clinical trials. Arthritis Rheumatol. 2015 Oct;67(10):2601-10. doi: 10.1002/art.39235. PMID 26097225
- [Background] Goncalves B, Ambrosio C, Serra S, Alves F, Gil-Agostinho A, Caseiro-Alves F. US-guided interventional joint procedures in patients with rheumatic diseases--when and how we do it? Eur J Radiol. 2011 Sep;79(3):407-14. doi: 10.1016/j.ejrad.2010.04.001. Epub 2010 Jun 4. PMID 20554144
- [Background] Andersen M, Ellegaard K, Hebsgaard JB, Christensen R, Torp-Pedersen S, Kvist PH, Soe N, Romer J, Vendel N, Bartels EM, Danneskiold-Samsoe B, Bliddal H. Ultrasound colour Doppler is associated with synovial pathology in biopsies from hand joints in rheumatoid arthritis patients: a cross-sectional study. Ann Rheum Dis. 2014 Apr;73(4):678-83. doi: 10.1136/annrheumdis-2012-202669. Epub 2013 Mar 8. PMID 23475981
- [Background] Sitt JC, Griffith JF, Wong P. Ultrasound-guided synovial biopsy. Br J Radiol. 2016;89(1057):20150363. doi: 10.1259/bjr.20150363. Epub 2015 Nov 2. PMID 26581578